CLINICAL TRIAL: NCT02226497
Title: Integrating a Telemonitoring Device Into the Outpatient Management of Adult Patients Following Intensive Chemotherapy for MDS and Non-APL AML: A Randomized Pilot Study
Brief Title: Telemonitoring Device in Managing Outpatient Care of Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia After Intensive Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 9105; NCI-2014-01680 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHCRC #9105; 9105 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-08-21; First posted 2014-08-27 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (standard outpatient supportive care) (Active Comparator): Patients receive standard outpatient supportive care after completion of chemotherapy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Supportive Care
- Arm II (home telemonitoring device) (Experimental): Patients receive standard outpatient supportive care as in Arm I and use the home telemonitoring device for the duration of chemotherapy-induced cytopenia (up to 3-4 weeks).
  Interventions: Device: Health Telemonitoring; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Supportive Care

INTERVENTIONS:
Device: Health Telemonitoring — Use home telemonitoring device
  Arms: Arm II (home telemonitoring device)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Supportive Care — Receive standard outpatient supportive care
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This randomized pilot clinical trial studies a home telemonitoring device in managing the care of patients with myelodysplastic syndrome or acute myeloid leukemia after they are discharged from the hospital following chemotherapy. After treatment and hospital discharge, patients typically need extensive care to deal with the side effects of chemotherapy, keep up with medications, and obtain medical assistance. A home telemonitoring device would allow patients to monitor vital signs, symptoms, and use of medications, communicate with healthcare providers, and access educational material. A telemonitoring device may allow patients to be managed more effectively than standard outpatient care after being discharged from the hospital.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of home telemonitoring for adult patients following intensive induction, re-induction/salvage, or consolidation chemotherapy for myelodysplastic syndrome (MDS) or non-acute promyelocytic leukemia (APL) acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To estimate the impact of the telemonitoring intervention on mortality, duration of hospital stay, use of emergency services, visits to primary care physicians and to specialists, home visits, and telephone calls ("health care resource utilization").

II. To evaluate the telemonitoring procedure in economic terms compared to usual care through a cost-effectiveness analysis.

III. To estimate the impact on the quality of life of study participating.

IV. To assess the degree of satisfaction of the patients/caregivers and health care professionals with the telemonitoring intervention.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (CONTROL): Patients receive standard outpatient supportive care after completion of chemotherapy.

ARM II (INTERVENTION): Patients receive standard outpatient supportive care as in Arm I and use the home telemonitoring device for the duration of chemotherapy-induced cytopenia (up to 3-4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS or AML other than APL with t(15;17)(q22;q12), (promyelocytic leukemia[PML]/retinoic acid receptor [RAR]), or variants according to the 2008 World Health Organization (WHO) classification
* Patient is currently undergoing AML-like intensive induction, re-induction/salvage, or consolidation chemotherapy, or planned to start such therapy within 1 week
* Willingness to have close follow-up and treatment at the Clinic at the Seattle Cancer Care Alliance (SCCA) or at a local facility; typically, patients will be seen at least 3 times per week as per standard practice, including at least once weekly at the SCCA
* Permanent or temporary housing available within a 60 minute (min) commute from the SCCA
* Available caregiver
* Willingness and ability to use the telemonitoring device
* Provision of written informed consent

Exclusion Criteria:

* Cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients willing to use the in-home telemonitoring device | Up to 4 weeks
  Exploratory, descriptive and observational methods will be used to determine enrollment and retention issues in AML/MDS patients who are discharged early after intensive chemotherapy.
Success of data transmission | Up to 4 weeks
  Exploratory, descriptive, and observational methods will be used to determine the ability to remotely monitor this patient population.

SECONDARY OUTCOMES:
Changes in patient conditions | Up to 4 weeks
  Researchers' ability to use the transmitted data to support patients in recognizing changes in their conditions and managing the changes or getting appropriate medical assistance will be estimated between study arms using exploratory, descriptive, and observational methods.
Degree of satisfaction of the patients/caregivers with the telemonitoring intervention | Up to 4 weeks (at end of study period)
  Exploratory, descriptive, and observational methods will be used to estimate differences between the study arms.
Degree of satisfaction of health care professionals with the telemonitoring intervention | Up to 4 weeks (at end of study period)
  Exploratory, descriptive, and observational methods will be used to estimate differences between the study arms.
Quality of life (QOL) as assessed by the M.D. Anderson Symptom Inventory Core items and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 | Up to 4 weeks (at end of study period)
  Exploratory, descriptive, and observational methods will be used to estimate in the impact of the telemonitoring intervention on QOL.
Percentage of returned surveys | Up to 4 weeks
  Percentage of returned surveys will be measured as a feasibility outcome.
Mortality | Up to 4 weeks
  The impact of the telemonitoring intervention on mortality compared to the control group will be estimated.
Health care resource utilization | Up to 4 weeks
  Descriptive and observational methods will be used to estimate the impact of the telemonitoring intervention with regard to health care resource utilization, and data on rehospitalization (frequency, duration, resource use, and need for intensive care unit-level care).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Halpern, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States